CLINICAL TRIAL: NCT06428084
Title: Comparative Efficacy of Dexamethasone - Ondansetron Versus Dexamethasone - Haloperidol in Reducing Postoperative Nausea and Vomiting After Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: Comparative Efficacy of Dexamethasone - Ondansetron Versus Dexamethasone - Haloperidol in Reducing PONV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AN-202405.01
Record Dates: First submitted 2024-05-16; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Laparoscopic Cholecystectomy
MeSH Terms: interventions — Ondansetron; Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ondansetron (Active Comparator): 19 participants in group O received 4 mg of ondansetron intravenously.
  Interventions: Drug: Ondansetron
- Haloperidol (Active Comparator): 19 participants in group H received 1 mg of Haloperidol intravenously.
  Interventions: Drug: Haloperidol

INTERVENTIONS:
Drug: Ondansetron — 4 mg of ondansetron intravenously
  Arms: Ondansetron
Drug: Haloperidol — 1 mg of Haloperidol intravenously
  Arms: Haloperidol

SUMMARY:
Nausea and vomiting following laparoscopic cholecystectomy remain common, with occurrence rates of 40-70% during the initial 24 hours post-operation. The underlying mechanisms of postoperative nausea and vomiting engage five distinct neurotransmitter receptors. Consequently, employing a combination of antiemetics from diverse classes that target various receptors for effective prevention is advised. Ondansetron's antiemetic properties derive from its ability to inhibit serotonin receptors, whereas Haloperidol targets dopamine receptors, and Dexamethasone reduces prostaglandin production.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) are also known as the little problem interpreted as a seemingly less significant complication but lead to increased morbidity, longer hospital stays, increased medical costs, and diminished patient satisfaction with healthcare services. These symptoms are reported more frequently than postoperative pain, making its prevention as important as postoperative pain management. In laparoscopic cholecystectomy, the occurrence of PONV can range from 40 - 70%, which is higher than the 33 - 49% observed in other types of surgeries under general anesthesia within the first 24 hours post-procedure. The mechanism of PONV is complex, involving multiple neurotransmitters. Targeted neurotransmitter receptors in the action of antiemetic drugs include muscarinic-1-acetylcholine (M1), dopamine-2 (D2), histamine-1 (H1), 5-Hydroxytryptamine-3-serotonin (5HT3), and neurokinin1-substance P (NK1) receptors. Based on this, the prevention of postoperative nausea and vomiting is recommended using a combination of various groups of antiemetics that work on different receptors. Studies have shown that combining different antiemetic classes is more effective than using a single agent. A meta-analysis study stated that dexamethasone, ondansetron, and droperidol are the most used types of antiemetics alone or in combination. Dexamethasone with a 5HT3 antagonist such as ondansetron is the most used antiemetic combination. Another viable option includes dexamethasone with Butypherone group drugs, such as droperidol, which acts as a D2 antagonist. However, droperidol was subject to FDA black box warnings in 2003 due to its association with arrhythmias caused by QT interval prolongation. Subsequent research has suggested haloperidol, another Butypherone group drug, as a safer alternative to droperidol.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic cholecystectomy
* aged 18 - 65 years
* ASA physical status 1 and 2
* Apfel score ≥2

Exclusion Criteria:

* a history of allergies
* routine use of antipsychotic drugs, steroids, antihistamines, and antiemetics before surgery
* cardiac rhythm disorders
* elevated liver enzyme levels (SGOT/SGPT) ≥5 times upper limit normal
* BMI ≥35 kg/m2

Dropout Criteria:

* if they experienced hypotension, defined as systolic blood pressure below 90 mmHg or mean arterial pressure (MAP) below 60 mmHg, or a decrease in systolic blood pressure and/or MAP greater than 20% from baseline for a duration exceeding two minutes, surgical procedures extending >3 hours, and any alterations in the planned surgical intervention.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Nausea and Vomiting Score | 24 hours post-operation
  Score 0 (No nausea, no vomiting); Score 1 (Nausea present, no vomiting); Score 2 (Nausea present, vomiting present); Score 3 (Vomiting >2 episodes in 30 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Dian Mardiani, M.D, Principal Investigator — Faculty of Medicine Universitas Padjadjaran Bandung
Locations (1):
- Hasan Sadikin General Hospital, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No